CLINICAL TRIAL: NCT02531789
Title: Procedure Outcome Predictor (POP) Using the Complement Cascade
Acronym: CPOP
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1011/115491
Record Dates: First submitted 2015-08-05; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Surgical Procedure Outcomes
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: 45 patients receiving elective colorectal surgery
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — C3, C4, CRP, and the dilution marker total IgG, together with C3dg, TCC and Bb will be measured over a high-sampling frequency time course t=-1 (admission), 0 (induction), 2,4,8,16, 24, 36 and 48 hours.

SUMMARY:
Current post-operative monitoring of patient recovery consists measuring two blood markers C-reactive protein (CRP) and White Blood Cell Count (WBC). However, these are slow to respond to the onset of infection. However, monitoring the absolute levels of the proteins in the three pathways of the complement cascade should provide a faster and better predictor of patient recovery. The investigators propose a pilot trial to measure concentrations of Complement Cascade (CC) activation biomarkers in the blood over a time course around operations of major abdomino-pelvic surgery involving a bowel resection. Further, analysis of the differential CC pathway activation should identify the onset of recovery complications before clinical symptoms present and potentially identify the causes allowing the clinicians to target therapies.

DETAILED DESCRIPTION:
The proposed study is a pilot study on a cohort of participants recruited from routine elective colorectal surgery at RD&E. The pilot trial will collect blood over a time course for a patient to record blood plasma levels of Complement proteins peri-operatively from admission to discharge. The assay schedule is detailed in Table 1 below. The trial will perform additional CC activation tests on routine blood samples taken during the patient's stay in hospital. In addition 4 trial samples will be taken at time intervals that will capture the impulse response of the patient's CC. Sample analysis will be performed in parallel in the clinical chemistry laboratory for laboratory for assays of CRP and the complement proteins C3 and C4. The additional trial assays will be performed on the MSD platform on loan for the period of the trial.

Table 1Blood Sample Assay Schedule Time Point Time of Test Routine Test Additional Trial Test Trial Assays Day Timings 0 t = -1 Pre-admission clinic CONSENT ROUTINE CRP, LFTs, FBC, Amylase, Coag, G&S C4, C5, IgG C3dg, C4d, Bb, TCC, t =-1 day 2 Pre-operatively t = 0 Under anaesthesia Trial Sample NO.1 C4, C5, IgG C3dg, C4d, Bb, TCC, CRP t = 0 9:30 hrs 3 t =1 hr Under anaesthesia Knife-to-skin plus 30 mins Trial Sample NO.2 C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 10.30 hrs 4 t = 2 - 4 hrs immediately post surgery ROUTINE C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 1330hrs (equivalent to t +4hrs) 5 t = 8 hrs Trial Sample NO. 3 C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 17:30 hrs 6 t = 12 hrs Trial sample NO. 4 C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 21:30 hrs 7 t = 24 hrs ROUTINE C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 09:30 hrs 8 t = 36 hrs ROUTINE C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 21:30 hrs 9 t = 48 hrs

Some Patients Discharged

Complications Develop ROUTINE C4, C5, IgG C3dg, C4d, Bb, TCC, CRP t = x1 Routine Tests as these occur C4, C5, IgG C3dg, C4d, Bb, TCC, CRP t = x2 Routine tests as these occur C4, C5, IgG C3dg, C4d, Bb, TCC, CRP 10 Discharge

The assays deployed for the pilot trial the current biomarkers of C activation panel are C3dg, C4d, Bb, TCC and the acute phase marker, CRP. The TCC assay has been designed in Cardiff (by Prof Morgan a collaborator of Prof Shaw) and the investigators have extensive experience in the design of C protein assays. For the target biomarkers antibodies to neo-antigens that are revealed post enzymatic cleavage or complex formation will be used as capture antibodies on the surface of the MSD platform. The C proteins are then detected with polyclonal antibodies provided by Prof Morgan in Cardiff and labelled with a ruthenium tagged antibody. Whole EDTA-stabilised plasma is then incubated in the 96-well format; all 5 assays, including calibration curves, are run simultaneously. Electroluminescence from the ruthenium complex is collected and quantified automatically. Absolute measurements of C proteins will be performed using standardised fully activated serum which contains a constant amount of activation products from all complement pathways. The serum is available through Prof Morgan's collaboration with the 'Complement Standardization Group'. C activation relative to this standard can then be determined. This work will lead to an array of C activation markers that will be tested against the patient cohort. This array including some of the other pathway markers may ultimately become the basis of a routine clinical test.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery list of pelvic oncology surgeons

Exclusion Criteria:

* Unable/unwilling to provide informed consent
* Pregnant women
* Under 18 years of age
* Pre-existing active infection
* Diabetic
* Inflammatory bowel disorders
* Immunosuppressed
* Immunosuppression or steroid treatment within the last 12 months
* Learning disability or mental health problems
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients receiving elective colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the Complement Activation with descriptive statistics to establish the size of an effect for a larger prospective cohort study | 5 days
  The study will determine Complement Cascade activation for a cohort of 45 patients receiving elective colorectal surgery. C3, C4, CRP, and the dilution marker total IgG, together with C3dg, TCC and Bb will be measured over a high-sampling frequency time course t=-1 (admission), 0 (induction), 2,4,8,16, 24, 36 and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Shaw, PhD, Principal Investigator — University of Exeter